CLINICAL TRIAL: NCT00142025
Title: Randomised, Placebo Controlled, Double Blind, Parallel Group 3-Months Study of Oxcarbazepine Efficacy in Asthma Therapy
Brief Title: Study of Efficacy of Oxcarbazepine in Therapy of Bronchial Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre of Chinese Medicine, Georgia (Other)
Collaborators: Rea Rehabilitation Centre, Georgia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP-0501-OC-0302
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Bronchial Asthma
Keywords: Bronchial asthma; Oxcarbazepine; Antiepileptic drug; Efficacy
MeSH Terms: conditions — Asthma | interventions — Oxcarbazepine

INTERVENTIONS:
Drug: Oxcarbazepine

SUMMARY:
The purpose of this study is to determine whether antiepileptic drug oxcarbazepine is effective in the treatment of chronic asthma.

DETAILED DESCRIPTION:
Effective therapy of asthma still remains quite serious problem. According GINA definition, asthma is an inflammatory disorder. Consequently, modern pharmacotherapy of asthma provides wide use of anti-inflammatory drugs. But asthma also is a paroxysmal disorder: many specialists and even some guidelines underline paroxysmal clinical picture of asthma. Besides this, according to some authors, neurogenic inflammation may play important role in asthma mechanism. But some other neurogenic inflammatory paroxysmal disorders exist, and they are migraine and trigeminal neuralgia. Some antiepileptic drugs, like carbamazepine and valproate, are very effective in therapy of migraine and trigeminal neuralgia - more than in 80% of cases. If bronchial asthma also is paroxysmal inflammatory disease, like migraine and trigeminal neuralgia, it is possible that some antiepileptic drugs also are very effective in asthma therapy.

We performed a double-blind, placebo-controlled 3-month trial for evaluation of oxcarbazepine efficacy in therapy of bronchial asthma. Oxcarbazepine is antiepileptic drug of new generation, produced by Novartis, and it is more effective and safe derivative of well-known antiepileptic drug carbamazepine.

Comparison: Patients received investigational drug in addition to their usual routine antiasthmatic treatment, compared to patients received placebo in addition to their usual routine antiasthmatic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Bronchial asthma has been known at least for 1 year
* Absence of long-term remissions of asthma (lasting more than 1 month)
* Poorly controlled asthma, due to various reasons
* Non-smokers

Exclusion Criteria:

* Presence of concomitant severe diseases
* Allergy or adverse reactions to carbamazepine or oxcarbazepine
* Abnormal baseline haematology, blood chemistry or urinalysis
* Current use of long-acting beta-agonists
* Age younger than 16 years old
* Long-term history of smoking
* Pregnancy or lactating

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55
Dates: Start 2001-09; Study Completion 2002-03

PRIMARY OUTCOMES:
At 3 months of treatment: Change from baseline of the FEV1 and PEFR (also %predicted); Number of patients without asthma symptoms

SECONDARY OUTCOMES:
At 3 months of treatment: FEV1 before and after salbutamol inhalation; Difference in PEF pm-am (in %); The daily (daytime and night-time) symptoms scores; % of symptom free days during the treatment period; Use of other antiasthmatic medication

CONTACTS AND LOCATIONS:
Overall Officials: Merab Lomia, MD, PhD, Principal Investigator — "Rea" Rehabilitation Centre.; Manana Tchaia, MD, Study Director — Centre of Chinese Medicine; Tamara Tchelidze, MD, Study Chair — CRO Evidence

REFERENCES:
- See also: Website of Neuroasthma Group — http://www.asthma.ge
- See also: Bronchial asthma as neurogenic paroxysmal inflammatory disease: a randomized trial with carbamazepine — http://www.ncbi.nlm.nih.gov/pubmed/16597501?ordinalpos=2&itool=EntrezSystem2.PEntrez.Pubmed.Pubmed_ResultsPanel.Pubmed_DefaultReportPanel.Pubmed_RVDocSum